CLINICAL TRIAL: NCT05360719
Title: Integrated Tele-exercise for Individuals With SCI: Physical, Psychological, and Social Responses With Spinal Cord Injury
Brief Title: Integrated Tele-exercise for Individuals With Spinal Cord Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: The Craig H. Neilsen Foundation (Other); Pennsylvania Department of Health (Other Government)
Responsible Party: Principal Investigator, Margaret A. Finley, Associate Professor, Principal Investigator, Drexel University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHNF865512-PADoH
Record Dates: First submitted 2022-04-13; First posted 2022-05-04 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury
Keywords: physical activity; group online exercise
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: waitlist control repeated measures
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor collecting data will be masked to group (wait list control vs immediate group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Tele-exercise Class (Experimental): Volunteers will be asked to participate in the group online exercise class 2 times per week for 8 weeks. Each activity session will last about 60 minutes and will focus on mind-body practices, tailored to physical and emotional needs of individuals with SCI. Class will be taught by a physical therapist who is an experienced community exercise instructor. Class will be co-led by a person who is living with SCI (one of our community partners). Classes will take place over a secure virtual platform (Zoom). Before beginning and after completion of the program, participants will be asked to participate in small group interviews to share expectations and experiences of the study
  Interventions: Behavioral: Group tele-exercise
- Waitlist Control (Other): The waitlist control group will complete all quantitative measures as a baseline (baseline-control) and will be instructed to continue their activities as usual, with measures obtained again at 8-weeks (post-control/pre-program). Following the initial 8-week baseline, each waitlist group will participate in pre-intervention semi-structured interview or small focus group with the post-control measures as pre-intervention assessment. They will join the tele-exercise intervention with all measures at 8-weeks (post-intervention) and with leisure time physical activity and quality of life assessed at 16-weeks following initiation of the program.
  Interventions: Behavioral: Group tele-exercise

INTERVENTIONS:
Behavioral: Group tele-exercise — This tele-exercise class will be tailored to the physical and emotional needs of individuals with SCI based on results of our feasibility study, the initial emergent themes from qualitative data collection in this study, and input from our co-leader with lived experience (examples: seated exercise to accommodate wheelchair users, active co-leader with SCI).The research clinician will lead the instruction of each class while our co-leader will model movements alongside her and offer tailored modifications as needed. Each 45-minute class provides a comprehensive fitness experience to maximize functional independence and improve global physical activity engagement. Elements incorporated into each class session include a collective check-in and breathing meditation, postural control, trunk and shoulder strength, cardiovascular fitness, and body awareness.

SUMMARY:
The objective of this study is to examine the efficacy of an integrated, participant-centered tele-health physical activity program for individuals with SCI on psychological and social factors through a parallel mixed-methods design approach. We will examine changes in psychological (self-efficacy, self-esteem, exercise outcome expectations, depression, positive affect and well-being, quality of life) and social factors (participation and satisfaction with social roles and activities, activity engagement) following participation in an 8-week integrated group tele-exercise health and wellness physical activity program, with retention assessed at 8-weeks following completion (16 weeks from baseline). We will also complete small group interviews with all participants to understand participant experiences of, response to, and recommendations before and following participation in group tele-exercise program.

To date, there is extremely limited evidence for the efficacy of psychological and social well-being of remotely delivered community-based exercise to individuals with SCI. A pilot effectiveness trial of a tele-exercise health and wellness program will be conducted using a mixed methods design with a randomized waitlist control group. Quantitative and qualitative data collection is sequential in nature and other data are collected simultaneously. Individuals with SCI (living with injury 12 months or longer) will be recruited based on existing partnerships locally and nationally. To assess limited effectiveness, we aim to enroll 35 individuals with SCI. Recruitment of these participants will stem from the investigator's ongoing community partnership with local and national partners. The tele-exercise health & wellness program will consist of virtual group class, twice per week, intended to generate physical confidence and strength for individuals living with SCI. Each session will be co-led with by an individual living with SCI.

DETAILED DESCRIPTION:
Physical activity participation directly impacts the body function and structures of individuals living with spinal cord injury (SCI). Physical inactivity can initiate and exacerbate secondary conditions that individuals with SCI are predisposed to including pressure sores, urinary tract infections, sleep disorders, and chronic pain. Kinesiophobia, a symptom related to pain, addresses an excessive and often debilitating fear of physical movement and activity and is associated with reduced level of physical activity. Individuals with newly acquired SCI have shown elevated levels of kinesiophobia during inpatient rehabilitation which remained unchanged at one-year. Specific to this proposal, there are numerous psychosocial benefits for individuals with SCI who participate in physical activity. These include reduction of depression and negative mood, increased self-confidence, improved body image, and enhanced quality of life. Qualitative findings support these outcomes in individuals with SCI who reported that physical activity reduced depressive moods, facilitated optimism and positive outlook, and helped manage stress; thus enhancing overall psychological well-being and mental health. Engagement in physical activity is positively associated with social quality of life. Participation created larger social networks and increased social achievement. Nearly 80% of individuals with SCI indicate that physical activity is important and express interest in maintaining an active lifestyle. However, internal barriers such as motivation and negative perceptions of physical activity have a strong association with exercise participation. Physical and financial barriers including inaccessible facilities, transportation complications, and cost of equipment further limit physical activity participation. Our recent work has further elucidated that barriers to community-based exercise with SCI have been exacerbated by the isolation required to minimize deleterious effects of the COVID-19 pandemic. Psychological and social isolation is increased in individuals with disabilities compared to nondisabled peers. These internal and external barriers highlight health and community inclusion disparities for individuals with SCI. Community inclusion provides people living with SCI equal access and opportunity to healthy living.

While there are numerous psychological and social benefits of exercise for individuals living with SCI, nearly 50% of this population is physically inactive. Tele-interventions have the potential to enhance physical activity participation and community inclusion through reducing barriers such as transportation and cost while improving access for individuals with SCI. Telehealth, or internet-based healthcare services, improve social support and increase cost-effectiveness as compared to standard of care practices. Telehealth has been cited as a successful strategy to mitigate SCI-related healthcare disparities and chronic health condition management. For example, telehealth is an effective intervention to manage pressure ulcer development in SCI. However, these findings are limited to case-based examination of healthcare provider clinical services. Evidence to support tele-interventions that also impact social engagement, such as group tele-exercise, is lacking. One small case-series demonstrated that participants with SCI valued group tele-exercise as a tool to overcome barriers to physical activity participation. Our study will provide evidence of the effectiveness of a community-based tele-exercise intervention for individuals with SCI to promote psychosocial well-being along with enhanced physical activity engagement.

This pragmatic effectiveness study will use a parallel, mixed methods, wait-list control group design. In order to more rigorously investigate the effectiveness of the tele-exercise intervention on psychological and social wellbeing, a subset of participants (n=10) will serve as controls through a waitlist control approach. To achieve this control group, following informed consent, the initial 20 participants will be randomized to immediate intervention group or waitlist control group, with the final 12 participants in the immediate intervention group. As the group tele-exercise intervention encourages participant interaction, the randomization will be in clusters of 6-10 participants. The immediate intervention group will participate in the pre-intervention a semi-structured interview or small focus group and quantitative measures will be obtained. They will participate in the tele-exercise intervention biweekly for 8 weeks with all measures (qualitative and quantitative) obtained at 8-weeks (post-intervention), with leisure time physical activity and quality of life assessed at 16-weeks following initiation of the program. The waitlist control group will complete all quantitative measures as a baseline (baseline-control) and will be instructed to continue their activities as usual, with measures obtained again at 8-weeks (post-control/pre-program). Following the initial 8-week baseline, each waitlist group will participate in pre-intervention semi-structured interview or small focus group with the post-control measures as pre-intervention assessment. They will join the tele-exercise intervention with all measures at 8-weeks (post-intervention) and with leisure time physical activity and quality of life assessed at 16-weeks following initiation of the program. All participants will be provided a logbook with instructions to document physical activity, reflections and associated emotions and behaviors.

ELIGIBILITY:
Inclusion Criteria:

* report a complete or incomplete SCI of ASIA grade A, B, C, or D
* living with injury at least 12 months
* self-reported ability to elevate shoulder 25% motion
* self-report being between 18-75 years of age
* self report not currently receiving structured rehabilitation,
* cleared by screen by ACSM guidelines for participation
* Internet access to participate in virtual classes

Exclusion Criteria:

* absolute contraindications as identified by ACSM21
* self-report previous hospitalization within a month
* self report active pressure ulcer
* self report recent osteoporotic fracture
* self-report uncorrectable vision loss,
* self report preexisting neurological conditions other than SCI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in narrative responses from focus group interviews at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  Semi-structured interviews or small tele-focus groups of 3-5 individuals that will take 60 minutes
Change in quality of life rating on the Subjective Quality of Life Questionnaire (SQoL) at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  This questionnaire is a global measure of subjective perception of QoL. The scale is a Likert-type scale measuring satisfaction with life as a whole: Participants are asked to take everything in their life into account and rate it on an ordinal scale from 1 (life is very distressing; it's hard to imagine how it could get much worse) to 7 (life is great; it's hard to imagine how it could get much better). Test-retest reliability is high (91% agreement), and this questionnaire is validated with the SCI population.
Change in pain interference on the Spinal Cord Injury Quality of Life - Measurement System-Pain Interference Short Form at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Pain Interference short form is comprised of 10 items, asking participants to rate their pain interference on an ordinal scale from 1 (not at all) to 5 (very much) where a higher sum score represents greater pain interference over the previous 7 days.
Change in pain behavior on the Spinal Cord Injury Quality of Life Measurement System-Pain Behavior Short Form at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Pain Behavior short form is comprised of 7 items, asking participants to rate their pain behavior on an ordinal scale from 1 (never) to 5 (always) for questions 1-3 and from 1 (had no pain) to 6 (always) in questions 4-7 where a higher sum score represents greater pain behavior over the previous 7 days.
Change in self-esteem on the Spinal Cord Injury Quality of Life Measurement System-Self-Esteem Short Form at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Self-Esteem short form is comprised of 8 items, asking participants to rate their pain behavior on an ordinal scale from 1 (never) to 5 (always) where a higher sum score represents decreased self-esteem with SCI.
Change in depression on the Spinal Cord Injury Quality of Life Measurement System-Depression Short Form at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Depression short form is comprised of 10 items, asking participants to rate their depressive symptoms on an ordinal scale from 1 (never) to 5 (always) where a higher sum score represents increased despair and/or loss of interest in things with SCI.
Change in resilience on the Spinal Cord Injury Quality of Life Measurement System-Resilience Short Form at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Resilience short form is comprised of 8 items, asking participants to rate their pain behavior on an ordinal scale from 1 (never) to 5 (always) where a higher sum score represents increased resilience with SCI.
Change in positive affect and well-being on the Spinal Cord Injury Quality of Life Measurement System-Positive Affect and Wellbeing Short Form at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Positive Affect and Wellbeing short form is comprised of 10 items, asking participants to rate their overall sense of purpose, wellbeing, and life satisfaction on an ordinal scale from 1 (never) to 5 (always) where a higher sum score represents increased positive affect and wellbeing with SCI.
Change in participation in social roles on the Spinal Cord Injury Quality of Life Measurement System-Participation in Social Roles and Activities Short Form at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Participation in Social Roles and Activities short form is comprised of 10 items, asking participants to rate their current involvement in social roles on an ordinal scale from 1 (never) to 5 (always) where a higher sum score represents increased participation in social roles and activities with SCI.
Change in satisfaction with social roles on the Spinal Cord Injury Quality of Life Measurement System-Satisfaction with Social Roles and Activities Short Form at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Participation in Social Roles and Activities short form is comprised of 10 items, asking participants to rate their current involvement in social roles on an ordinal scale from 1 (not at all) to 5 (very much) where a higher sum score represents increased satisfaction with social roles and activities with SCI.
Change in sleep disturbance on the General Sleep Disturbance Scale at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  The GSDS is a 21-item scale was designed to evaluate the incidence and nature of sleep disturbances. Questions pertain to a variety of general sleep issues, including problems initiating sleep, waking up during sleep, waking too early from sleep, quality of sleep, quantity of sleep, fatigue and alertness at work, and the use of substances to induce sleep. Internal consistency for the full scale has been shown to be 0.88. The GSDS queries respondents regarding the frequency with which they've experienced certain sleep difficulties within the previous week. Respondents use an eight-point, Likert-type scale ranging from 0 (meaning "never") to 7 ("every day") to respond to each item where higher sum score represents increased general sleep disturbance.
Change in exercise self-efficacy on the Exercise Self-Efficacy Scale at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  This self-report measures the construct of self-efficacy, or personal beliefs in one's capabilities relating to exercise participation in individuals with SCI. Self-efficacy is cited as the most critical personal factor to behavior change. This outcome demonstrates reliability and high internal consistency. Respondents answer using a 4-point Likert-type scale ranging from 1 (not at all true) to 4 (exactly true) to respond to 10-items where higher sum score represents increased exercise self-efficacy with SCI.
Change in exercise outcome expectations on the Multidimensional Outcome Expectations for Exercise (MOESS) at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  The Multidimensional Outcome Expectations for Exercise Scale (MOEES). This self-report measure addresses physical, social, and self-evaluative components of outcome expectations, another critical element needed for health behavior change.This tool also demonstrates high internal consistency and validity. Respondents answer using a 5-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree) to respond to 15-items where higher sum score represents increased positive exercise outcome expectations.
Change in leisure time physical activity behavior on the Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) at Week 8 | Pre-Program (0 weeks) and Post-Program (8 weeks)
  The Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) is an SCI-specific, self-report measure of leisure-time physical activity that assesses minutes of mild, moderate, and heavy intensity leisure-time physical activity performed over the previous 7-days. Test-retest reliability and criterion validity of the LTPAQ-SCI has been established. Total number of exercise minutes over the previous 7-days is calculated.

SECONDARY OUTCOMES:
Accelerometry | One time collection during intervention
  A subset of participants (n=5-10) will receive a wearable activity monitor to be used during a class within weeks 6-8 of the tele-exercise class program. Physical activity monitoring will be performed using one accelerometer (ActiGraph GT3X+) placed on the nondominant wrist of the participant. Participant instruction on use of the accelerometer with occur remotely. Participants can contact the team if they have any issues using the device. Accelerometry data for a one to two 45-minute exercise sessions per participant will be recorded and transformed into minutes of moderate-vigorous physical activity. This will be completed using open-source MIMS unit algorithms based on individually developed thresholds.
Change in quality of life rating on the Subjective Quality of Life Questionnaire (SQoL) at Week 16 | Post-Program (8 weeks) and Retention (16 weeks)
  This questionnaire is a global measure of subjective perception of QoL. The scale is a Likert-type scale measuring satisfaction with life as a whole: Participants are asked to take everything in their life into account and rate it on an ordinal scale from 1 (life is very distressing; it's hard to imagine how it could get much worse) to 7 (life is great; it's hard to imagine how it could get much better). Test-retest reliability is high (91% agreement), and this questionnaire is validated with the SCI population.
Change in leisure time physical activity behavior on the Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) at Week 16 | Post-Program (8 weeks) and Retention (16 weeks)
  The Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) is an SCI-specific, self-report measure of leisure-time physical activity that assesses minutes of mild, moderate, and heavy intensity leisure-time physical activity performed over the previous 7-days. Test-retest reliability and criterion validity of the LTPAQ-SCI has been established. Total number of exercise minutes over the previous 7-days is calculated.
Change in exercise self-efficacy on the Exercise Self-Efficacy Scale at Week 16 | Post-Program (8 weeks) and Retention (16 weeks)
  This self-report measures the construct of self-efficacy, or personal beliefs in one's capabilities relating to exercise participation in individuals with SCI. Self-efficacy is cited as the most critical personal factor to behavior change. This outcome demonstrates reliability and high internal consistency. Respondents answer using a 4-point Likert-type scale ranging from 1 (not at all true) to 4 (exactly true) to respond to 10-items where higher sum score represents increased exercise self-efficacy with SCI.
Change in exercise outcome expectations on the Multidimensional Outcome Expectations for Exercise (MOESS) at Week 16 | Post-Program (8 weeks) and Retention (16 weeks)
  The Multidimensional Outcome Expectations for Exercise Scale (MOEES). This self-report measure addresses physical, social, and self-evaluative components of outcome expectations, another critical element needed for health behavior change.This tool also demonstrates high internal consistency and validity. Respondents answer using a 5-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree) to respond to 15-items where higher sum score represents increased positive exercise outcome expectations.
Change in quality of life rating on the Subjective Quality of Life Questionnaire (SQoL) from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  This questionnaire is a global measure of subjective perception of QoL. The scale is a Likert-type scale measuring satisfaction with life as a whole: Participants are asked to take everything in their life into account and rate it on an ordinal scale from 1 (life is very distressing; it's hard to imagine how it could get much worse) to 7 (life is great; it's hard to imagine how it could get much better). Test-retest reliability is high (91% agreement), and this questionnaire is validated with the SCI population.
Change in pain interference on the Spinal Cord Injury Quality of Life - Measurement System-Pain Interference Short Form from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Pain Interference short form is comprised of 10 items, asking participants to rate their pain interference on an ordinal scale from 1 (not at all) to 5 (very much) where a higher sum score represents greater pain interference over the previous 7 days.
Change in pain behavior on the Spinal Cord Injury Quality of Life Measurement System-Pain Behavior Short Form from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Pain Behavior short form is comprised of 7 items, asking participants to rate their pain behavior on an ordinal scale from 1 (never) to 5 (always) for questions 1-3 and from 1 (had no pain) to 6 (always) in questions 4-7 where a higher sum score represents greater pain behavior over the previous 7 days.
Change in self-esteem on the Spinal Cord Injury Quality of Life Measurement System-Self-Esteem Short Form from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Self-Esteem short form is comprised of 8 items, asking participants to rate their pain behavior on an ordinal scale from 1 (never) to 5 (always) where a higher sum score represents decreased self-esteem with SCI.
Change in depression on the Spinal Cord Injury Quality of Life Measurement System-Depression Short Form from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Depression short form is comprised of 10 items, asking participants to rate their depressive symptoms on an ordinal scale from 1 (never) to 5 (always) where a higher sum score represents increased despair and/or loss of interest in things with SCI.
Change in resilience on the Spinal Cord Injury Quality of Life Measurement System-Resilience Short Form from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Resilience short form is comprised of 8 items, asking participants to rate their pain behavior on an ordinal scale from 1 (never) to 5 (always) where a higher sum score represents increased resilience with SCI.
Change in positive affect and well-being on the Spinal Cord Injury Quality of Life Measurement System-Positive Affect and Wellbeing Short Form from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Positive Affect and Wellbeing short form is comprised of 10 items, asking participants to rate their overall sense of purpose, wellbeing, and life satisfaction on an ordinal scale from 1 (never) to 5 (always) where a higher sum score represents increased positive affect and wellbeing with SCI.
Change in participation in social roles on the Spinal Cord Injury Quality of Life Measurement System-Participation in Social Roles and Activities Short Form from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Participation in Social Roles and Activities short form is comprised of 10 items, asking participants to rate their current involvement in social roles on an ordinal scale from 1 (never) to 5 (always) where a higher sum score represents increased participation in social roles and activities with SCI.
Change in satisfaction with social roles on the Spinal Cord Injury Quality of Life Measurement System-Satisfaction with Social Roles and Activities Short Form from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories of recovery and outcomes of interventions/rehabilitation. The measure demonstrates excellent test-retest reliability (ICC = 0.84). The Participation in Social Roles and Activities short form is comprised of 10 items, asking participants to rate their current involvement in social roles on an ordinal scale from 1 (not at all) to 5 (very much) where a higher sum score represents increased satisfaction with social roles and activities with SCI.
Change in sleep disturbance on the General Sleep Disturbance Scale from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  The GSDS is a 21-item scale was designed to evaluate the incidence and nature of sleep disturbances. Questions pertain to a variety of general sleep issues, including problems initiating sleep, waking up during sleep, waking too early from sleep, quality of sleep, quantity of sleep, fatigue and alertness at work, and the use of substances to induce sleep. Internal consistency for the full scale has been shown to be 0.88. The GSDS queries respondents regarding the frequency with which they've experienced certain sleep difficulties within the previous week. Respondents use an eight-point, Likert-type scale ranging from 0 (meaning "never") to 7 ("every day") to respond to each item where higher sum score represents increased general sleep disturbance.
Change in exercise self-efficacy on the Exercise Self-Efficacy Scale from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  This self-report measures the construct of self-efficacy, or personal beliefs in one's capabilities relating to exercise participation in individuals with SCI. Self-efficacy is cited as the most critical personal factor to behavior change. This outcome demonstrates reliability and high internal consistency. Respondents answer using a 4-point Likert-type scale ranging from 1 (not at all true) to 4 (exactly true) to respond to 10-items where higher sum score represents increased exercise self-efficacy with SCI.
Change in exercise outcome expectations on the Multidimensional Outcome Expectations for Exercise (MOESS) from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  The Multidimensional Outcome Expectations for Exercise Scale (MOEES). This self-report measure addresses physical, social, and self-evaluative components of outcome expectations, another critical element needed for health behavior change.This tool also demonstrates high internal consistency and validity. Respondents answer using a 5-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree) to respond to 15-items where higher sum score represents increased positive exercise outcome expectations.
Change in leisure time physical activity behavior on the Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) from baseline to pre-program (Waitlist control group only) | Baseline to Pre-Program
  The Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) is an SCI-specific, self-report measure of leisure-time physical activity that assesses minutes of mild, moderate, and heavy intensity leisure-time physical activity performed over the previous 7-days. Test-retest reliability and criterion validity of the LTPAQ-SCI has been established. Total number of exercise minutes over the previous 7-days is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Finley, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baehr LA, Hiremath SV, Bruneau M Jr, Chiarello LA, Kaimal G, Newton R, Finley M. Effect of Tele-exercise to Promote Empowered Movement for Individuals With Spinal Cord Injury (TEEMS) Program on Physical Activity Determinants and Behavior: A Mixed Methods Assessment. Arch Phys Med Rehabil. 2024 Jan;105(1):101-111. doi: 10.1016/j.apmr.2023.08.019. Epub 2023 Sep 9. PMID 37678447